CLINICAL TRIAL: NCT00143728
Title: A Randomized Study to Evaluate Virologic Response Following Discontinuation vs. no Discontinuation of 3TC in Patients Who Are Infected With HIV With Previously Documented Reduced Susceptibility to 3TC and Who Have Adequate Virologic Suppression on Combination Antiretroviral Therapy
Brief Title: 3TC or No 3TC for HIV With 3TC Resistance
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment.
Sponsor: University of British Columbia (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Dr. Julio Montaner, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03-0051; CTN 189
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Lamivudine

INTERVENTIONS:
Drug: Lamivudine — See Detailed Description.

SUMMARY:
The purpose of this study is to compare the effects of continuing or discontinuing 3TC treatment in the presence of HIV virus with 3TC resistance for persons who are on a regimen including least three other anti-HIV drugs. The overall aim is to determine whether continuing 3TC is of benefit in HIV-positive persons who have already shown resistance to this drug.

ELIGIBILITY:
Inclusion Criteria:

* Be HIV positive
* Be at least 18 years old.
* Currently receiving 3TC for HIV infection in conjunction with at least three other antiretroviral drugs. Must have started this regimen at least three months prior to starting this study.
* A plasma viral load of less than 50 copies/mL on at least two occasions (measured at least 28 days apart immediately prior to screening).
* Evidence of resistance to 3TC

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Hepatitis B surface antigen (HbsAg) positive at time of screening or with the previous year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2004-01; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Virologic failure (VL above 50 copies/ml) on two consecutive dates, at least two weeks apart, in the absence of concurrent acute illness or recent immunization during the first 24 weeks. | 24 weeks

SECONDARY OUTCOMES:
Percent and absolute change in viral load from baseline to week 24 and week 48. | 48 weeks
Change in CD4 count in both absolute number and percentage from baseline to week 24 and week 48. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julio Montaner, MD, Principal Investigator — University of British Columbia/Providence Health Care
Locations (9):
- Canada (9):
  - Downtown IDC, Vancouver, British Columbia
  - Cool Aid Community Health Centre, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Haven Program, Greater Sudbury, Ontario
  - McMaster University, Hamilton, Ontario
  - Maple Leaf Clinic, Toronto, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Centre Hospitalier de l'université de Laval, Ste-Foy, Quebec